CLINICAL TRIAL: NCT07395739
Title: A Phase I, Randomized, Double-blinded, Positive-Controlled Clinical Trial to Assess the Safety and Immunogenicity of the Group B Meningococcal OMV Vaccine (DX-104) in Adults Aged 18 to 50 Years
Brief Title: A Phase I Clinical Trial to Assess the Safety and Immunogenicity of DX-104
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yuguan Biotech Co., Ltd.（Delonix Bioworks) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C-104-003
Record Dates: First submitted 2026-01-23; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neisseria Meningitidis Serogroup B
MeSH Terms: interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Because the investigational vaccine and the comparator vaccine have distinct visual appearances, the care provider administering the vaccination cannot remain blinded, while participants and other investigators will maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DX-104 (Experimental): Participants in this arm will receive three doses of DX-104 at Months 0, 1, and 6.
  Interventions: Biological: Group B Meningococcal OMV Vaccine
- Bexsero® (Active Comparator): Participants in this arm will receive three doses of Bexsero® at Months 0, 1, and 6.
  Interventions: Biological: Bexsero®

INTERVENTIONS:
Biological: Bexsero® — Intramuscular injection; 0.5ml/pre-filled syringe. Administer the vaccine according to the 0, 1, 6-month schedule.
  Arms: Bexsero®
Biological: Group B Meningococcal OMV Vaccine — Intramuscular injection; 0.5ml/vial. Administer the vaccine according to the 0, 1, 6-month schedule.
  Other Names: DX-104
  Arms: DX-104

SUMMARY:
A randomized, double-blinded, positive-controlled clinical trial will be conducted to observe the safety and immunogenicity of DX-104 in adults 18 to 50 years of age.

DETAILED DESCRIPTION:
A total of 30 healthy participants will be enrolled and randomized (2:1) to receive DX-104 or Bexsero® (multicomponent meningococcal group B vaccine). Participants in both the DX-104 and Bexsero® groups will receive three doses of intramuscular vaccination at Months 0, 1, and 6.

After all participants have completed the 6-month safety and immunogenicity observations following full vaccination, the trial will be concluded.

ELIGIBILITY:
Inclusion Criteria

1. Healthy male or female participants aged 18 to 50 years (inclusive) at the time of screening, who can provide valid legal identification.
2. Willing and able to give written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
3. Willing and able to comply with all study procedures and available for the entire duration of the study follow-up.
4. Participants must have a Body Mass Index (BMI) between ≥18.0 and ≤32.0 kg/m2 at screening.
5. For female participants at least 1 of the following conditions must apply:

   i) Is not of childbearing potential (WONCBP), defined as surgically sterile (hysterectomy, bilateral salpingectomy, tubal ligation or bilateral oophorectomy - verbal confirmation through medical history review acceptable) or postmenopausal (no menses for 12 months and confirmed by FSH level ≥40 mIU/mL); or ii) Is of childbearing potential (WOCBP), has negative pregnancy tests at screening and prior to the first vaccination, and agrees to: Practice true abstinence (where this is consistent with their usual lifestyle); or Use a highly effective method of contraception consistently from signing the consent form until 6 months after the last vaccination. Highly effective contraception includes hormonal contraception (oral, injected, implanted or transdermal) plus use of a condom, placement of an intrauterine device (IUD) or intrauterine system (IUS) plus use of a condom, or a vasectomized male partner (performed at least 6 months prior) who has been documented to no longer produce sperm - verbal confirmation through medical history review acceptable; or iii) Are in an exclusively same-sex relationship. iv) In addition, pre-menopausal women must agree not to donate their ova from signing the consent form until at 6 months after the last vaccination.
6. Females should not be currently breastfeeding, and should not breastfeed for the duration of the study.
7. Male participants are able to participate if they:

   i) Practice true abstinence (where this is consistent with their usual lifestyle); or ii) Are surgically sterilized (performed at least 6 months prior and documented to no longer produce sperm - verbal confirmation through medical history review acceptable); or iii) If their female partner is a WOCBP, the male participant must use a condom and the WOCBP female partner must use a highly effective contraception method (i.e. established use of hormonal contraception started at least 30 days prior to Day 0/Visit 1; or placement or an IUD), from screening and for 6 months after the last vaccination; or iv) Are in an exclusively same sex relationship. v) In addition, non-sterile males must agree not to donate their sperm from signing the consent form until 6 months after the last vaccination.

Exclusion Criteria

1. Oral temperature >37.5°C at screening or prior to vaccination* 2. Previous vaccination with any Group B meningococcal vaccine (including GSK's Bexsero® or Pfizer's Trumenba®) or a history of invasive disease caused by Neisseria meningitidis.

3. Individuals with abnormal findings in pre-vaccination laboratory tests, vital signs, physical examination, or electrocardiogram (ECG) that are deemed clinically significant by the Investigator or delegate. * 4. Known allergy or hypersensitivity to any component of the investigational vaccine, or a history of severe allergic reactions (including, but not limited to: anaphylaxis, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, Arthus reaction, dyspnea, angioneurotic edema, etc.).

5. Administration of any live-attenuated vaccine within 14 days (inclusive) prior to vaccination, or any other subunit, inactivated, or recombinant protein vaccine within 7 days (inclusive) before vaccination.* 6. Acute illness or exacerbation of a chronic illness within 3 days prior to vaccination.* 7. Use of antipyretics, analgesics, or anti-allergy medications within 24 hours prior to vaccination. * 8. Long-term use of immunomodulators within 3 months prior to screening (e.g., systemic corticosteroids for ≥14 days at a dose of ≥2 mg/kg/day or ≥20 mg/day of prednisone or equivalent), or planned use during the study period. Note: Topical preparations (e.g., ointments, eye drops, inhalers, nasal sprays) are permitted.

9. Receipt of blood products and/or immunoglobulins within 3 months prior to vaccination, or planned administration during the study period.* 10. Participants who have donated or lost more than 450 mL of blood within 30 days before the screening visit. * 11. Participants with any severe underlying disease, congenital malformation, or ongoing medical condition that, in the judgment of the investigator or delegate, may pose a risk to the participant or interfere with the conduct, safety, or scientific validity of the trial. This includes, but is not limited to: active or latent tuberculosis (Mycobacterium tuberculosis), symptomatic or poorly controlled respiratory diseases such as asthma or chronic bronchitis, Down syndrome, thalassemia, heart disease, kidney disease, autoimmune disorders, atopic predisposition, Guillain-Barré syndrome, current skin diseases, etc.

12. Participants with encephalopathy, uncontrolled epilepsy, convulsions, other progressive neurological disorders, or a significant personal history of psychiatric disorders.

13. Contraindications to intramuscular injection, including, but not limitedto: diagnosed thrombocytopenia, any coagulation disorder, or current treatment with anticoagulants. 14. Asplenia, functional asplenia, or splenectomy due to any reason. 15. Planned relocation from the local area before trial completion or prolonged absences scheduled during the trial visit periods.

16. Participation in another clinical trial involving an investigational or unregistered product (drug, vaccine, device, etc.) within 30 days prior to vaccination, or planned participation in any other clinical trial before the completion of this study.* 17. Positive test for hepatitis C virus (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) or syphilis at screening.

18. Participants with skin conditions that in the opinion of the investigator or delegate may interfere with the assessment of local adverse reactions (e.g., tattoos at the injection site, psoriasis, plaques affecting the skin in the deltoid area, etc.).

19. Any other condition which, in the opinion of the Investigator or delegate, may compromise the assessment of the trial objectives.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
To assess the overall safety of DX-104 | Through study completion, an average of 1 year.
  1. The incidence and severity of any AEs within 30 days after each vaccination.
  2. The incidence and severity of any AEs within 30 minutes after each vaccination.
  3. The incidence and severity of any solicited local and systemic AEs within 7 days after each vaccination.
  4. The incidence and severity of any unsolicited AEs within 30 days after each vaccination.
  5. The occurrence of clinically significant laboratory abnormalities on Day 3 after each vaccination.
  6. The incidence of any serious adverse events (SAEs) from the first vaccination until 6 months after the last vaccination.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Geometric mean titers (GMTs) of serum bactericidal antibody against meningococcal B strains, as measured by serum bactericidal assays using human complement (hSBA), at Day 30 following each vaccination and at 6 months after the last vaccination.
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Geometric mean-fold rise (GMFR) relative to baseline of serum bactericidal antibody against meningococcal B strains, as measured by serum bactericidal assays using human complement (hSBA), at Day 30 following each vaccination and at 6 months after the last vaccination.
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Seroconversion rate (SCR) of serum bactericidal antibody against meningococcal B strains, as measured by serum bactericidal assays using human complement (hSBA), at Day 30 following each vaccination and at 6 months after the last vaccination.
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Geometric mean titers (GMTs) of Immunoglobulin G (IgG) against meningococcal B strains, as measured by ELISA, at Day 30 following each vaccination and at 6 months after the last vaccination.
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Geometric mean-fold rise (GMFR) relative to baseline of Immunoglobulin G (IgG) against meningococcal B strains, as measured by ELISA, at Day 30 following each vaccination and at 6 months after the last vaccination.
To evaluate the immunogenicity of DX-104 | Through study completion, an average of 1 year.
  Seroconversion rate (SCR) of Immunoglobulin G (IgG) against meningococcal B strains, as measured by ELISA, at Day 30 following each vaccination and at 6 months after the last vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Early Phase Limited, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided